CLINICAL TRIAL: NCT01237860
Title: Evaluation of the Safety and Performance of the NESS L300 Plus System
Acronym: L300Plus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bioness Inc (Industry)
Collaborators: Bioness Neuromodulation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 001 Rev 04
Record Dates: First submitted 2010-11-08; First posted 2010-11-10 (Estimated); Last update posted 2011-11-16 (Estimated); Status verified 2011-11

CONDITIONS: Foot Drop; Thigh Muscles Weakness (Hamstrings or Quadriceps); Upper Motor Neuron Injury or Disease
Keywords: Foot drop; Thigh muscle weakness; Upper Motor Neuron injury or disease
MeSH Terms: conditions — Peroneal Neuropathies; Disease | interventions — Drug Delivery Systems

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: NESS L300 Plus System — The patients will receive the device for daily use of six (6) weeks.
  Other Names: NESS L300; L300; L300 Plus

SUMMARY:
The study is designed to evaluate the safety and efficacy of using the L300 Plus as a neuroprosthesis device for walking in patients following an UMN injury or disease. The clinical study is proposed to determine the anticipated adverse event rate and treatment outcomes at the conclusion of the study.

DETAILED DESCRIPTION:
This is a prospective, one-center, single group, repeated measures, non inferiority study. Forty-five (45) subjects suffering from foot drop and thigh muscles weakness due to upper motor neuron injury or disease will be evaluated for this study. Each subject will be in the study for six weeks. Clinical benefits will be measured through an assessment of the gait performance. In particular it will test the hypothesis that the NESS L300 Plus System which involves foot drop correction with thigh muscles activation, may achieve walking enhancements not inferior to those gained from using a system that only corrects foot drop (i.e. NESS L300).

ELIGIBILITY:
Inclusion Criteria:

* Upper motor neuron lesion
* Thigh muscle weakness - hamstrings or quadriceps strength of less than 4/5 according to manual muscle testing
* Foot drop - toe drag during walking
* Lower limb spasticity - 0-4 according to the modified Ashworth scale
* Responsible mental state, able to follow multiple step directions
* Between 18 and 80 years old
* Available for participation in the study
* Able to understand and sign the informed consent form
* Able to walk independently or with an assistance device (e.g. cane, walker etc.) / spot guarding for at least 10 meters
* Sufficient response to electrical stimulation (visible muscle contractions in a seated or prone position of each designated muscle separately)

Exclusion Criteria:

* Subjects with a demand-type cardiac pacemaker, defibrillator or any electrical or metallic implant
* Cancerous lesion of lower limb, present or suspected
* Medical condition that prevents participation or would likely lead to inability to comply with the protocol [e.g.: congestive heart failure, patient receiving chemotherapy, uncontrolled epilepsy, etc]
* Severe cognitive impairment (MMSE<21)
* Severe neglect (Star cancellation test<30)
* Skin lesion at the site of the stimulation electrodes
* Change in bone-joint structures of the lower limb, such as contractures or deformations; fracture or dislocation, which would be adversely affected by motion from the stimulation
* Pregnancy
* Diagnosis of major depression or psychotic disorder
* Participation in another investigation that may directly or indirectly affect the study results
* Unable to tolerate electrical stimulation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2010-09; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Occurence of anticipated and unanticipated adverse events | Throughout the 6 weeks of the study
  The occurence of anticipated and unanticipated events will be documented at each scheduled evaluation. In addition, subjects will be instructed to report adverse events 24 hours per day during the study period.
Subject feedback regarding the safety of using the device | Week 6
  Patient feedback regarding the safety of using the device as reported during the study sessions and the completion of a satisfaction questionnaire will also be used to assess the system's safety.

SECONDARY OUTCOMES:
Temporal Gait Parameters of the 2 Minute Walk Test | Week 1 and Week 6
  This outcome measure includes the following: gait velocity, gait asymmetry, single limb support (percentage of the singe stance phase).
10 Meter Obstacle Course Walking Velocity | Week 1 and Week 6
  To imitate daily life situations, average gait speed will be also determine by measuring the time to walk 10m over an obstacle course, using the protocol in the Emory Functional Ambulation Profile.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Jacques Vatine, MD, Principal Investigator — Reuth Rehabilitation Hospital
Locations (1):
- Reuth Medical Center, Tel Aviv, Israel

REFERENCES:
- [Background] Bonita R, Solomon N, Broad JB. Prevalence of stroke and stroke-related disability. Estimates from the Auckland stroke studies. Stroke. 1997 Oct;28(10):1898-902. doi: 10.1161/01.str.28.10.1898. PMID 9341692
- [Background] Robbins SM, Houghton PE, Woodbury MG, Brown JL. The therapeutic effect of functional and transcutaneous electric stimulation on improving gait speed in stroke patients: a meta-analysis. Arch Phys Med Rehabil. 2006 Jun;87(6):853-9. doi: 10.1016/j.apmr.2006.02.026. PMID 16731222
- [Background] Glanz M, Klawansky S, Stason W, Berkey C, Chalmers TC. Functional electrostimulation in poststroke rehabilitation: a meta-analysis of the randomized controlled trials. Arch Phys Med Rehabil. 1996 Jun;77(6):549-53. doi: 10.1016/s0003-9993(96)90293-2. PMID 8831470
- [Background] Yan T, Hui-Chan CW, Li LS. Functional electrical stimulation improves motor recovery of the lower extremity and walking ability of subjects with first acute stroke: a randomized placebo-controlled trial. Stroke. 2005 Jan;36(1):80-5. doi: 10.1161/01.STR.0000149623.24906.63. Epub 2004 Nov 29. PMID 15569875
- [Background] Hausdorff JM, Ring H. Effects of a new radio frequency-controlled neuroprosthesis on gait symmetry and rhythmicity in patients with chronic hemiparesis. Am J Phys Med Rehabil. 2008 Jan;87(1):4-13. doi: 10.1097/PHM.0b013e31815e6680. PMID 18158427